CLINICAL TRIAL: NCT03347383
Title: Physician Initiated, Prospective, Non-randomized Belgian Multi-center Trial, Investigating the Safety and Efficacy of the Treatment With the LumINor DCB and The IvolutioN Stent of iVascular in TASC C and D Femoropopliteal Atherosclerotic Disease
Brief Title: Clinical Trial Investigating the Combination Therapy With Luminor DCB and iVolution Stent in TASC C and D Femoropopliteal Lesions
Acronym: TINTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID3-20170628
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Stents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy DCB + stent (Experimental): Patients treated with the Luminor DCB and the iVolution stent
  Interventions: Device: Combination therapy DCB + stent

INTERVENTIONS:
Device: Combination therapy DCB + stent — Patients will be treated with the Luminor DCB and iVolution stent

SUMMARY:
The T.I.N.T.I.N. study investigates the safety and efficacy of the combination therapy with the Luminor drug coated balloon (DCB) and the iVolution stent in the treatment of TASC C and D femoropopliteal lesions. An expected total of 100 patients will be treated in the scope of this study. The lesion is located within the native superficial femoral artery and/or the popliteal artery. Prior to dilatation with the Luminor DCB, pre-dilatation with the Oceanus balloon is mandatory. After dilatation with the Luminor DCB, stenting with the iVolution stent need to be performed. Post-dilatation can be performed according to the physician's discretion. Patients will be invited for a follow-up visit at 1, 6, 12, 24, 36, 48 and 60 month post-procedure. The primary efficacy endpoint of the study is defined as the freedom from clinically-driven target lesion revascularization (TLR) at 12 months. Secondary endpoints include primary patency rate at 6 and 12 months, freedom from clinically-driven TLR at 6, 24, 36, 48 and 60 months, clinical success at 1, 6, 12, 24, 36, 48 and 60 months and freedom from serious adverse events at pre-discharge, 1, 6, 12, 24, 36, 48 and 60 months follow-up.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate, in a controlled setting, the long-term safety and efficacy of the combination therapy with the Luminor DCB and the iVolution stent post CE-certification and according to the indications of the Instructions for use (IFU) with focus on the treatment of TASC C and D femoropopliteal atherosclerotic lesions.

Patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should also be geographically stable, willing and able to cooperate in this clinical study and remain available for long-term follow-up. A patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following tests and clinical data will be collected: informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of chronic limb ischemia (Rutherford category) and resting ankle-brachial index (ABI).

During the procedure, the vascular access can be achieved to the investigator's standard clinical practice. After successful lesion passage, diagnostic angiography of the lesion area and distal run-off is performed and angiographic measurements (vessel diameter, percentage stenosis and lesion length) are collected. All inflow-limiting lesion will be treated according to the investigators standard clinical practice before treatment of the target lesion. Pre-dilatation of the target lesion is mandatory with the Oceanus balloon. After pre-dilatation, a least one Luminor DCB will be inflated and at least 1 iVolution stent will be deployed at the target lesion. At the physician's discretion, post-dilatation can be performed. No other adjunctive therapies (atherectomy, laser) are allowed. The complete femoropopliteal vasculature should be treated in one single session, staged interventions are not allowed. All outflow-limiting lesions must be treated according to the hospital treatment standard.

The regular follow-ups are necessary to monitor the condition of the patient and the procedure. Patients will be invited for a follow-up visit at 1, 6, 12, 24, 36, 48 and 60 months after the index procedure. The 24, 36, 48 and 60 month follow-up can be conducted via a phone call. The following data will be collected during these follow-up visit: medication record, physical examination, rutherford categorization, ABI and color flow doppler ultrasound.

ELIGIBILITY:
General inclusion criteria:

* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life expectancy of at least 12 months
* Prior to enrolment, the guidewire has crossed target lesion
* Patient is eligible for treatment with the Luminor Paclitaxel-Eluting Peripheral Balloon Dilatation Catheter and the iVolution stent
* Male, infertile female or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure

Angiographic inclusion criteria

* De novo and post-percutaneous transluminal angioplasty (PTA) restenotic lesions located in the femoropopliteal arteries suitable for endovascular therapy
* The target lesion is located within the native femoropopliteal artery
* The length of the target lesion is ≥ 150mm and considered as TASC C or D lesion according to the TASC II classification.
* The target lesion has angiographic evidence of stenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* Target vessel diameter visually estimated is >4mm and <6.5 mm
* There is angiographic evidence of at least one-vessel-runoff to the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention

Exclusion Criteria:

* Patient refusing treatment
* Presence of a stent in the target lesion that was placed during a previous procedure
* Untreated flow-limiting inflow lesions
* Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Patients with uncorrected bleeding disorders
* Aneurysm located at the level of the superficial femoral artery/popliteal artery
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (severe chronic obstructive pulmonary disease, metastatic malignancy, dementia, etc.) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Use of thrombectomy, atherectomy or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, M.D., Study Director — ID3 Medical
Locations (9):
- Belgium (9):
  - O.L.V. Hospital, Aalst
  - Z.N.A., Antwerp
  - Imelda Hospital, Bonheiden
  - Sint-Jozefkliniek, Bornem
  - A.Z. Sint-Blasius, Dendermonde
  - H. Hartziekenhuis, Lier
  - AZ Damiaan, Ostend
  - R.Z. Heilig Hart, Tienen
  - AZ Jan Portaels, Vilvoorde

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 study subjects were enrolled in a period of 14 months, between September 2017 and October 2018.
Pre-assignment Details: All enrolled patients were treated with the study device.
Groups:
- Combination Therapy DCB + Stent: A total of 100 study subjects were enrolled in a period of 14 months, between September 2017 and October 2018.
  Combination therapy DCB + stent: Patients were treated with the Luminor DCB and iVolution stent.
  Patients were followed for 5 years.
Period: Overall Study
Arm/Group | Combination Therapy DCB + Stent
Started | 100
Completed | 49
Not Completed | 51
Not completed — Death | 39
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 100
Nicotine abuse [Count of Participants; unit: Participants]
  Former | 22
  current | 48
  never | 30
Hypertension [Count of Participants; unit: Participants] | 73
Diabetes [Count of Participants; unit: Participants] | 37
Hypercholesterolemia [Count of Participants; unit: Participants] | 63
Obesity [Count of Participants; unit: Participants] | 32
History of peripheral artery intervention [Count of Participants; unit: Participants] | 40
History of coronary intervention [Count of Participants; unit: Participants] | 23
History of cerebrovascular intervention [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Clinically-driven TLR at 12 Months
Description: Freedom from clinically-driven TLR at 12 months: defined as a repeated intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at the respective time points
Time Frame: 12-month
Population: At twelve month, 5 patients had a TLR, 7 patients died, 1 withdrew his consent and 1 patient was lost-to-follow-up
Measure: Number; unit: participants
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
participants | 5

2. Secondary Outcome: Primary Patency Rate
Description: Primary patency rate at 6-,12-month follow-up; defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.5) at the target lesion and without TLR within the time of procedure and the given follow-ups
Time Frame: 6 and 12 months post-procedure
Measure: Number; unit: participants
Groups:
- Combination Therapy DCB + Stent at 6 Month: A total of 100 study subjects were enrolled in a period of 14 months, between September 2017 and October 2018.
  Combination therapy DCB + stent: Patients were treated with the Luminor DCB and iVolution stent.
  Patients were followed for 5 years.
Arm/Group | Combination Therapy DCB + Stent at 6 Month
Number analyzed (Participants) | 100
participants
  Number of patient who lost their Primary patency at 6 months | 7
  Number of patient who lost their Primary patency at 12 months | 8

3. Secondary Outcome: Technical Success
Description: Technical success: defined as the ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30%
Time Frame: Index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
Participants | 100

4. Secondary Outcome: Freedom From Clinically-driven TLR
Description: Freedom from clinically-driven Target Lesion Revascularisation (CD-TLR) at 6-month, 2-, 3-, 4- and 5-year follow-up; TLR defined as a repeated intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at the respective time points
Time Frame: 6, 24, 36, 48 and 60 months post-procedure
Measure: Number; unit: participants
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
participants
  Number of patients with CD-TLR at 6 months | 1
  Number of patients with CD-TLR at 2 years | 10
  Number of patients with CD-TLR at 3 years | 17
  Number of patients with CD-TLR at 4 years | 20
  Number of patients with CD-TLR at 5 years | 25

5. Secondary Outcome: Clinical Success
Description: Clinical success at follow-up is defined as an improvement of Rutherford classification at 1-, 6-, 12-, 24-, 36-, 48- and 60-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months post-procedure
Population: Not all patients had a 1 to 60-month follow-up (e.g. missed visits, patients died, lost-to follow-up, ....) . As a result, not all 100 rutherford measurements were available for each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
Participants
  Number of patients whose RCC was improved compared to baseline at 1-month follow-up.: number analyzed (Participants) | 94
  Number of patients whose RCC was improved compared to baseline at 1-month follow-up. | 84
  Number of patients whose RCC was improved compared to baseline at 6-month follow-up.: number analyzed (Participants) | 85
  Number of patients whose RCC was improved compared to baseline at 6-month follow-up. | 79
  Number of patients whose RCC was improved compared to baseline at 12-month follow-up.: number analyzed (Participants) | 79
  Number of patients whose RCC was improved compared to baseline at 12-month follow-up. | 74
  Number of patients whose RCC was improved compared to baseline at 24-month follow-up.: number analyzed (Participants) | 59
  Number of patients whose RCC was improved compared to baseline at 24-month follow-up. | 56
  Number of patients whose RCC was improved compared to baseline at 36-month follow-up.: number analyzed (Participants) | 48
  Number of patients whose RCC was improved compared to baseline at 36-month follow-up. | 47
  Number of patients whose RCC was improved compared to baseline at 48-month follow-up.: number analyzed (Participants) | 40
  Number of patients whose RCC was improved compared to baseline at 48-month follow-up. | 39
  Number of patients whose RCC was improved compared to baseline at 60-month follow-up.: number analyzed (Participants) | 28
  Number of patients whose RCC was improved compared to baseline at 60-month follow-up. | 25

6. Secondary Outcome: Serious Adverse Events (SAEs)
Description: Serious adverse events as defined per ISO 14155:2011
Time Frame: up to 60 months post-procedure
Measure: Number; unit: serious adverse events
Arm/Group | Combination Therapy DCB + Stent
Number analyzed (Participants) | 100
serious adverse events | 226

ADVERSE EVENTS:
Time Frame: 5 years post procedure
Groups:
- Combination Therapy DCB + Stent: At the time of this 60-month follow-up report, there were 295 adverse events. 226 events were serious adverse events (SAEs). Of the 295 events, 61 were indicated as mild, 125 as moderate and 109 as severe. Forty-seven were study lesion related, 39 events were device related and 25 events were procedure related. The device and procedure related events were classified as highly probable, probable or unlikely related. Thirty-nine subjects died in this 60-month follow-up period, from which none of the causes of death were procedure or device related. All device and procedure related events reported during this period are considered anticipated.
Arm/Group | Combination Therapy DCB + Stent
All-Cause Mortality (participants affected / at risk) | 39/100
Serious Adverse Events (participants affected / at risk) | 80/100
Other Adverse Events (participants affected / at risk) | 44/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy DCB + Stent (N=100)
Anemia (Blood and lymphatic system disorders) | 2 (2)
CVA (Vascular disorders) | 2 (2)
CVA resulted in death (Vascular disorders) | 2 (2)
Other (Blood and lymphatic system disorders) | 4 (4)
Post-transplant lymphoproliferative disorder resulted in death (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
CABG (Cardiac disorders) | 1 (1)
Cardiac arrest resulted in death (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 4 (4)
Heart failure resulted in death (Cardiac disorders) | 3 (3)
Other (Cardiac disorders) | 1 (1)
Difficult metabolic control of DM type 1 (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Carcinoma resulted in death (Gastrointestinal disorders) | 1 (1)
Colon carcinoma (Gastrointestinal disorders) | 1 (1)
Colon polyps (Gastrointestinal disorders) | 2 (2)
Gastro-intestinal bleeding resulted in death (Gastrointestinal disorders) | 1 (1)
Obstruction (Gastrointestinal disorders) | 2 (2)
Other (Gastrointestinal disorders) | 3 (3)
Deterioration of general health resulted in death (General disorders) | 10 (10)
Deterioration of general health (General disorders) | 3 (3)
Organ failure resulted in death (General disorders) | 1 (1)
Other (General disorders) | 7 (10)
Sepsis (General disorders) | 2 (2)
Sepsis resulted in death (General disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
COVID infection resulted in death (Infections and infestations) | 3 (3)
Foot wound (Infections and infestations) | 4 (4)
Fracture (Musculoskeletal and connective tissue disorders) | 5 (5)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Other (Musculoskeletal and connective tissue disorders) | 3 (5)
Large intracranial bleeding resulted in death (Blood and lymphatic system disorders) | 1 (1)
Dementia resulted in death (Nervous system disorders) | 1 (1)
Epileptic seizure resulted in death (Nervous system disorders) | 1 (1)
Other (Nervous system disorders) | 2 (4)
Stroke resulted in death (Nervous system disorders) | 2 (2)
Vertigo (Nervous system disorders) | 1 (1)
AV fistula procedure (Renal and urinary disorders) | 3 (3)
Renal insufficiency (Renal and urinary disorders) | 3 (5)
Infection (Renal and urinary disorders) | 2 (2)
Kidney insufficiency resulted in death (Renal and urinary disorders) | 1 (1)
Chronic lung disease with emphysema resulted in death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Long embolism resulting in death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung cancer resulting in death (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia resulted in death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure resulted in death (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tumour (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Foot wound (Skin and subcutaneous tissue disorders) | 8 (14)
Aneurysm (Vascular disorders) | 4 (4)
Arterial stenosis/occlusion (Vascular disorders) | 39 (83)
Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy DCB + Stent (N=100)
burn wound (Skin and subcutaneous tissue disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Other (Blood and lymphatic system disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 3 (3)
Cardiac decompensation (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Inflammation (Gastrointestinal disorders) | 1 (1)
Infection (Gastrointestinal disorders) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1)
Dizzines (General disorders) | 1 (1)
Gout (General disorders) | 1 (1)
Other (General disorders) | 1 (2)
Arthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Inflammation (Musculoskeletal and connective tissue disorders) | 2 (2)
Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inflammation (Skin and subcutaneous tissue disorders) | 2 (2)
Wound (Skin and subcutaneous tissue disorders) | 3 (3)
Edema (Skin and subcutaneous tissue disorders) | 4 (4)
Arterial stenosis/occlusion (Vascular disorders) | 20 (21)
Pseudoaneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03347383/Prot_SAP_000.pdf